CLINICAL TRIAL: NCT05857033
Title: Effectiveness of Cold Vibratory Stimuli on Pain Perception Governing Infiltration Anesthesia in the Maxillary Arch in Children: a Randomized Controlled Clinical Trial
Brief Title: Cold Vibratory Stimuli on Pain Perception Governing Infiltration Anesthesia in in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0568-12/2022
Record Dates: First submitted 2023-04-26; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia, Local
Keywords: Dental injection; Palatal injection; Indirect palatal injection

STUDY DESIGN:
Intervention Model Description: The Participants will be randomly and equally allocated into 2 groups with 2 subgroups each
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Direct local anesthesia with Buzzy (Experimental)
  Interventions: Other: Buccal and direct palatal injection with the aid of Buzzy
- Indirect local anesthesia with Buzzy (Experimental)
  Interventions: Other: Buccal and indirect palatal injection with the aid of Buzzy
- Direct local anesthesia (Active Comparator)
  Interventions: Other: Buccal and direct palatal injection without Buzzy
- Indirect local anesthesia (Active Comparator)
  Interventions: Other: Buccal and indirect palatal injection without Buzzy

INTERVENTIONS:
Other: Buccal and direct palatal injection with the aid of Buzzy — Children are assigned to local anesthesia after using the Buzzy vibration unit extraorally for 2 minutes using buccal and direct palatal injection
  Arms: Direct local anesthesia with Buzzy
Other: Buccal and indirect palatal injection with the aid of Buzzy — Children are assigned to local anesthesia after using the Buzzy vibration unit extraorally for 2 minutes using buccal and indirect palatal injection
  Arms: Indirect local anesthesia with Buzzy
Other: Buccal and direct palatal injection without Buzzy — Children are assigned to local anesthesia after using topical analgesic gel (benzocaine 20%) intraorally for 1 minute using buccal and direct palatal injection
  Arms: Direct local anesthesia
Other: Buccal and indirect palatal injection without Buzzy — Children are assigned to local anesthesia after using topical analgesic gel (benzocaine 20%) intraorally for 1 minute using buccal and indirect palatal injection
  Arms: Indirect local anesthesia

SUMMARY:
Local anesthesia injections are sometimes painful, resulting in antagonistic cooperation, fear, and anxiety in children. This study aims to investigate the effectiveness of vibratory and cold stimulation before the injection to reduce pain. Purpose of the study: Evaluate the effectiveness of Buzzy® in pain reduction during local anesthesia administration compared to the traditional topical anesthetic gel in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are in need of extraction of maxillary posterior teeth.
* Children free of any systemic disease or special health care needs (ASA I).
* Children with no learning disabilities.
* Positive or definitely positive behavior during preoperative assessments according to the Frankl Scale.
* Patients whose parents will give consent to participate.

Exclusion Criteria:

* Having active sites of pathosis in the area of injection that could affect the anesthetic assessment.
* Signs of reversible pulpitis.
* Restorable tooth.
* Patients allergic to local anesthesia or having a family history of allergy to local anesthesia.
* Patients with acute oral or facial infection (swelling and/or cellulites )

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | Baseline and up to 1 hour
  Visual Analogue Scale is used and it ranges from 0 to 10. the ''0'' point indicates ''no pain'' and ''10'' point indicates the worst possible pain.
Change in child's behavior | During the procedure
  Sound, eye,motor (SEM) scale is used. it assess child's pain perception by observing discomfot levels on SEM during injections.
  Total scores for SEM range from 0 to 9 based on 0-3 score for each parameter. Score 0: Comfort Score 1: Mild disocomfort Score 2: Moderate discomfort Score 3: Severe discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Hambouta HM, Sharaf DA, Wahba NA. Effectiveness of cold vibratory stimuli on pain perception governing infiltration anesthesia in the maxillary arch in children: a randomized controlled clinical trial. BMC Oral Health. 2025 Jun 3;25(1):900. doi: 10.1186/s12903-025-06170-4. PMID 40462040